CLINICAL TRIAL: NCT03680430
Title: Phase II Study Evaluating Adaptive Radiation Therapy in Pre-operative or Exclusive Radiation Therapy for Limb Soft Tissues Sarcomas
Brief Title: Evaluation of Adaptive Radiation Therapy in Pre-operative or Exclusive Radiation Therapy for Limb Soft Tissues Sarcomas
Acronym: ADAPTO-SARC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADAPTO-SARC-IPC 2017-030
Record Dates: First submitted 2018-09-20; First posted 2018-09-21 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Sarcoma, Soft Tissue
Keywords: adaptive image guided radiation therapy; limb soft tissues sarcomas
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- limb soft tissue sarcoma (Experimental)
  Interventions: Radiation: Adaptive radiation therapy

INTERVENTIONS:
Radiation: Adaptive radiation therapy — Patients will be treated by preoperative or definitive radiotherapy for a limb STS, using an intensity-modulated conformal irradiation (with a static or dynamic technic), over 5 to 7 consecutive weeks. The total dose delivered will be of 50 Gray (preoperative RadioTherapy), or 60 to 70 Gray (exclusive RadioTherapy).

SUMMARY:
Soft tissue sarcomas (STS) is generally treated by surgery, followed or preceded by radiotherapy and chemotherapy. Preoperative irradiation has been shown to be effective in a randomized trial, and is often indicated in locally advanced Soft tissue sarcomas of the limbs, in order to reach R0 resection, or in case of rapid tumor growth despite first chemotherapy. For inoperable sarcomas, radiotherapy is an efficient palliative treatment, increasing local control.

Adaptive radiotherapy is defined as the set of procedures leading to the modification of a treatment plan based on the individual variations observed during irradiation. The place of this technique is increasing since the development of image-guided-radiotherapy allowing the visualization of daily variations in position, shape or volume of the tumor and organs at risk. Its implementation in current practice however remains limited because of the cumbersome processes involved (new delineation, new dose calculation, or even re-optimization) and resources to commit, especially in human time.

Irradiation of soft tissue sarcomas always begins with a planning CT scan, where the target-volumes and organ at risk are delineated, and dosimetric calculations are performed prior to radiotherapy initiation. During the radiotherapy, the variations leading to a mismatch between the planned dose and the dose delivered are multiple. These may be due to positioning errors or morphological changes in the patient (weight loss), or in the tumor or organs at risk (modifications in shape, size or position). The volume of soft tissue sarcomas changes also during radiotherapy (response, progression or pseudo- progression of the tumor).

However, to date, few data are available in the literature both on the volume variation of soft tissue sarcomas during preoperative radiotherapy, and on the interest of adaptive radiotherapy in the management of these tumors. It is therefore necessary to evaluate whether modifications of growth or macroscopic tumor volume are observed during the treatment, and to evaluate dosimetric impact on the target volume coverage that could impact the results of the treatment.

This a prospective multicentric phase II trial conducted to evaluate the interest of adaptive radiotherapy in the preoperative or exclusive management of limb sarcomas Patients will be treated by preoperative or definitive radiotherapy for a limb soft tissue sarcomas, using an intensity-modulated conformal irradiation (with a static or dynamic technic), over 5 to 7 consecutive weeks. The total dose delivered will be of 50 Gray (preoperative radiation therapy), or 60 to 70 Gray (exclusive radiation therapy). The delineation of growth or macroscopic tumor volume,clinical target volume, and planning target volume, as well as healthy surrounding tissues will be carried out in each of the centers, and under the responsibility of the radiotherapist, on The simulation CT-scan, used for dosimetry, and 3 CT scan performed on day 1 of radiotherapy (d1), at a dose of 30Gy (d30Gy) and 50Gy (d50GY). The dosimetric re-planning according to the variations of the volume of the planning target volume will be done in case of significant variation of the target volume according to de definition mentionned in the main and secondary objectives.

Main objective: The aim of this study is to evaluate the interest of adaptive radiotherapy in the preoperative or exclusive management of limb sarcomas.

This is the first prospective trial focused on the evaluation of the volume variation of soft tissue sarcomas during preoperative radiotherapy, and also on the interest of adaptive radiotherapy in the management of these tumors, whereas indications of preoperative and/or exclusive radiation therapy are very frequent.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have signed the written consent
* Age ≥ 18 years
* Patient with a diagnosis of sarcoma of the limbs (including buttock and shoulder)
* Treatment by preoperative or exclusive radiotherapy (more or less concomitant chemotherapy)
* Patient affiliated to the national "Social Security" regimen or beneficiary of this regimen

Exclusion Criteria:

* Patient with a diagnosis of sarcoma of the head and neck, retroperitoneum, trunk or abdomen
* Person in urgent situation, person of legal age subject to a measure of legal protection (major under guardianship, guardianship or court bail), or unable to express his / her consent
* Impossibility of submitting to the medical examination of the test for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2019-06-20 (Estimated); Primary Completion 2020-09-20 (Estimated); Study Completion 2020-09-20 (Estimated)

PRIMARY OUTCOMES:
Variations in growth or macroscopic tumor volume | 3 months
  proportion of patients with clinically significant variations in growth or macroscopic tumor volume. Will be considered clinically significant the following variations of more than 10%

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Paoli-Calmettes, Marseille, Bouches-du-Rhônes, France

IPD SHARING:
Plan to Share IPD: No